CLINICAL TRIAL: NCT01269450
Title: The Impact of Progesterone on the Risk of Preterm Birth Among Women With Second Trimester Bleeding. A Double Blind Placebo Controlled Trial
Brief Title: Progesterone and Second Trimester Bleeding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, Dr., HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0023-08-EMC
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Antepartum Bleeding; Preterm Birth
Keywords: second trimester vaginal bleeding; late abortion; preterm birth; progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Utrogestan (Active Comparator)
  Interventions: Drug: micronized progesterone 200 mg (Utrogestan)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: micronized progesterone 200 mg (Utrogestan) — micronized progesterone 200 mg (Utrogestan, company) as an intra-vaginal tablet once daily
  Arms: Utrogestan
Drug: placebo — placebo 200mg vaginal tablets
  Arms: placebo

SUMMARY:
Working hypothesis and aims:

To investigate whether progesterone treatment affects the incidence of preterm labor compared to placebo, among women with 2nd trimester bleeding.

The participants will be allocated through randomization to a study or control group. Women in the study group will receive micronized progesterone 200 mg (Utrogestan, company) with an intra-vaginal tablet once daily while the control group will receive placebo. Both women and medical staff will be blinded to group allocation. Treatment will commence on the day of inclusion to the study, but not before 16 weeks and will continue until 36 weeks gestation. Data will be collected after the conclusion of pregnancy regarding the maternal and neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Viable pregnancy
* Gestational age between 13 to 26 weeks
* Vaginal bleeding from uterine origin
* Singleton pregnancy
* Normal clotting tests
* Hemodynamically stable woman

Exclusion Criteria:

* Water leak
* Signs of preterm labor
* Fetal malformations incompatible with life
* Uterine malformations and other maternal conditions, i.e. liver disease, breast cancer, active thromboembolic state
* Past preterm birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Incidence of spontaneous preterm birth - before 37 weeks. | 3 years

SECONDARY OUTCOMES:
Maternal and fetal outcomes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: RAED SALIM, MD, Principal Investigator — HaEmek medical center affiliated to the Rappaport faculty of medicine, Technion, Haifa, Israel
Locations (3):
- Israel (3):
  - Emek medical center, Afula
  - dEP ob/gyn, Hillel Yaffe Medical Center., Hadera
  - Dep. OB/GYN, The Nazareth Hospital, E.M.M.S, Nazareth

REFERENCES:
- [Derived] Salim R, Hakim M, Zafran N, Nachum Z, Romano S, Garmi G. Double-blind randomized trial of progesterone to prevent preterm birth in second-trimester bleeding. Acta Obstet Gynecol Scand. 2019 Oct;98(10):1318-1325. doi: 10.1111/aogs.13641. Epub 2019 Jun 1. PMID 31087325